CLINICAL TRIAL: NCT03976895
Title: Effect of Prone Position on the Use of Non-invasive and Invasive Ventilation in Infants With Moderate to Severe Acute Bronchiolitis
Brief Title: Prone Position in Acute Bronchiolitis
Acronym: PROPOSITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0333
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Viral Bronchiolitis
Keywords: viral bronchiolitis; Prone position; high flow nasal cannula; noninvasive ventilation; Randomized controlled trial
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — Supine Position; Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine position (SP) (Other): Supine position (SP) combined with HFNC
  Interventions: Procedure: Supine position (SP)
- Prone position (PP) (Experimental): Prone position (SP) combined with HFNC
  Interventions: Procedure: Prone position (PP)

INTERVENTIONS:
Procedure: Supine position (SP) — Infants under high flow nasal cannula (HFNC) will be positioned in the supine position.
  Patients may be positioned temporarily in lateral position between periods of supine position to limit ventilatory disorders, as it is usually done in critical care units during bronchiolitis.
  Arms: Supine position (SP)
Procedure: Prone position (PP) — Infants under high flow nasal cannula (HFNC) will be placed in the prone position during at least 24 hours over the first 48 hours. The positioning will be standardized (chest on the bed plan and abdomen cleared) and children should be placed in the prone position immediately after randomization.
  Patients may be positioned temporarily in lateral position between periods of prone position to limit ventilatory disorders, as it is usually done in critical care units during bronchiolitis.
  Arms: Prone position (PP)

SUMMARY:
Acute viral bronchiolitis is the leading cause of community-acquired acute respiratory failure in developed countries (20 000 to 30 000 hospitalizations each year in France). Between 5% and 22% of these children are hospitalized in a critical care unit to benefit from a respiratory support.

Non-invasive ventilation, in particular the nasal Continuous Positive Airway Pressure (nCPAP), reduces the work of breathing in children with bronchiolitis and is associated with decreased morbidity and hospitalization costs compared with invasive ventilation. Nowadays, this technique is considered as the gold standard in the pediatric intensive care units (PICU) in France. High Flow Nasal Cannula (HFNC) has been proposed as an alternative to the nCPAP because of its better tolerance and simplicity of implementation. However, the proportion of failure remains high (35 to 50%), providing only a partial response to the care of these children, especially prior to the PICU.

In a physiological study (NCT02602678, article published), it has been demonstrated that prone position (PP) decrease, by almost 50%, the respiratory work of breathing and improve the respiratory mechanics in infants hospitalized in intensive care units for bronchiolitis.

Investigators hypothesize that prone position, during High Flow Nasal Cannula (HFNC), would significantly reduce the use of non-invasive ventilation (nCPAP and others) or invasive ventilation, as compared to supine position during HFNC, in infants with moderate to severe viral bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Infant under 6 months
* Hospitalized in critical care unit (continuous monitoring unit or intensive care unit)
* With a clinical diagnosis of acute viral bronchiolitis (criterion of the American Academy of Pediatrics 2014)
* m-WCAS score ≥ 3 and / or hypercapnic acidosis with pH <7.35 and pCO2> 50mmHg (6.7 kPa)
* Informed consent signed by at least one of the parents with oral consent of the other parent (and / or legal guardian) recorded in the medical file.

Exclusion Criteria:

* Infant admitted with criteria for invasive or non-invasive ventilation (hypercapnic acidosis with pH <7.25 without ventilatory support and/or hypoxia with impossibility of maintaining SpO2> 92% whatever the FiO2 and/or more than 3 significant apneas per hour and/or severe consciousness disorder)
* Patient already positioned in the prone position before randomization
* Significant comorbidities with a history of respiratory pathology (bronchodysplasia with ventilatory support), Ear Nose and Throat pathology (pharyngolaryngomalacia) or neuromuscular and / or hemodynamically significant congenital heart disease.
* Contraindication to Prone position : recent abdominal surgery (laparoschisis or omphalocele) or recent sternotomy
* Patient who is not affiliated (or does not benefit from) to a national social security system

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion of ventilated children in each of the 2 groups | 3 days
  Indications for the use of ventilation (invasive or non-invasive ventilation) will be standardized in both groups (based on the interregional protocol for the management of bronchiolitis):
  * Clinical aggravation defined by an increase ≥ 1 point of the m-WCAS score
  * Persistence of hypercapnic acidosis with pH ≤7.30 and pCO2≥ 8 kPa or FiO2> 60% under HFNC at 2 L/kg/min
  * More than 2 significant apneas per hour (apnea with desaturation <90% and / or bradycardia <90 / min)
  * Consciousness disorder
  Anytime over the first 3 days after inclusion

SECONDARY OUTCOMES:
Proportion of failure | 3 days
  Failure is defined as:
  * HFNC failure (composite failure criterion validated by an independent committee)
  * worsening of mWCAS score ≥ 1 point
  * hypercapnic acidosis (pH ≤7.30 and pCO2≥8kPa)
  * significant apnea (apnea with desaturation <90% and / or bradycardia <90/min)
  Anytime over the first 3 days after inclusion
Causes of failure | 3 days
  Failure is defined as:
  * HFNC failure (composite failure criterion validated by an independent committee)
  * worsening of mWCAS score ≥ 1 point
  * hypercapnic acidosis (pH ≤7.30 and pCO2≥8kPa)
  * significant apnea (apnea with desaturation <90% and / or bradycardia <90/min)
  Anytime over the first 3 days after inclusion
Duration of ventilation | maximum 3 months
  Duration of ventilation (high flow nasal cannula, invasive, non-invasive) in hours.
  This data will be collected at critical care unit discharge.
Length of stay | maximum 3 months
  Length of stay in days. This data will be collected at hospital discharge.
Oxygenation evaluation | 2 hours
  Evolution of FiO2 and SpO2/FiO2 ratio between inclusion and H2.
Oxygenation evaluation | 12 hours
  Evolution of FiO2 and SpO2/FiO2 ratio between inclusion and H12.
Oxygenation evaluation | 24 hours
  Evolution of FiO2 and SpO2/FiO2 ratio between inclusion and H24.
Tolerance evaluation | maximum 3 months
  Proportion of skin lesions, vomiting/regurgitation and exclusive enteral nutrition.
  This data will be collected at critical care unit discharge.
Variation EDIN score (Scale of pain and discomfort of the newborn) between inclusion and after 2 hours | 2 hours
  Scale ranges to 0 from 15 and is a combination of criteria:
  * Face: Relaxed=0 to Permanent tightness or prostrate face,frozen or purple face=3
  * Body: Relaxed=0 to Permanent agitation,tightness of extremities and stiffness of limbs or very poor and limited motor skills with fixed body=3
  * Sleep:Easily, extended and calm=0 to No sleep=3
  * Relationship:Smile to the angels,smile answer,attentive to the listening=0 to Refuses contact,no relationship possible,howl or moan without any stimulation=3
  * Comfort: Do not need comfort=0 to Inconsolable,desperate sucking=3
Evaluation of the feasibility of maintaining the position | 48 hours
  Proportion of children in the prone position repositioned definitively in the supine position before performing the cumulative 24 hours of prone position, cumulative hours of prone position in the first 48 hours

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Réanimation pédiatrique et unité de surveillance continue - Hôpital Femme Mère Enfant - Hospices Civils de Lyon, Bron
  - CHU de Caen, Service de réanimation et surveillance continue pédiatrique, Caen
  - CH CHAMBERY Unité de surveillance continue pédiatrique, Chambéry
  - CH CLERMONT FERRAND Service de réanimation néonatal et pédiatrique, CHU Estaing, Clermont-Ferrand
  - Hôpital d'Enfants CHU de Dijon Service de réanimation pédiatrique, Dijon
  - CH ANNECY GENEVOIS Unité de surveillance continue pédiatrique, Épagny
  - CH VILLEFRANCHE Service de pédiatrie néonatologie, Gleizé
  - CHU GRENOBLE Service de réanimation pédiatrique Hôpital Couple Enfant, La Tronche
  - CHU MONTPELLIER Service de réanimation pédiatrique, Montpellier
  - CHU Nantes Unité de surveillance continue pédiatrique Hôpital mère-enfant, Nantes
  - CHU LENVAL NICE Service de réanimation pédiatrique, Nice
  - Hôpital Necker Enfant Malade, Paris Service de Réanimation et surveillance continue médicochirurgicales, Paris
  - CHU SAINT-ETIENNE Service de réanimation pédiatrique, Saint-Priest-en-Jarez
  - Hôpital Hautepierre CHU de Strasbourg Service de réanimation pédiatrique spécialisée, Strasbourg
  - Hôpital Clocheville Service de réanimation pédiatrique et d'USC médico-chirurgicale CHRU Tours, Tours
  - CRHU Nancy Réanimation Pédiatrique Spécialisée, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No